CLINICAL TRIAL: NCT00110279
Title: Phase I Inpatient Study of the Safety and Immunogenicity of H9N2 (6-2) AA ca Reassortant (A/Chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca), a Live Attenuated Virus Vaccine Candidate for Prevention of Avian Influenza H9N2 Infection in the Event of a Pandemic (Study A)
Brief Title: Safety of and Immune Response to a Bird Flu Virus Vaccine (H9N2) in Healthy Adults (Study A)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Ruth Karron, MD, Center for Immunization Research, Johns Hopkins School of Public Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIR 211 (Study A); H.22.05.03.11.B2
Record Dates: First submitted 2005-05-05; First posted 2005-05-06 (Estimated); Last update posted 2008-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Influenza; Virus Diseases
Keywords: Bird Flu
MeSH Terms: conditions — Influenza, Human; Virus Diseases; Influenza in Birds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): One vaccination with H9N2 (6-2) AA ca Reassortant (A/chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca) vaccine at a dose of 10^7 TCID50 delivered by nose drops.
  Interventions: Biological: H9N2 (6-2) AA ca Reassortant (A/chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca)
- 2 (Experimental): One vaccination with H9N2 (6-2) AA ca Reassortant (A/chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca) vaccine at a dose of 10^7 TCID50 delivered by nose drops. This Arm will enroll 4 weeks after Arm 1. Enrolled volunteers must have participated in Arm 1.
  Interventions: Biological: H9N2 (6-2) AA ca Reassortant (A/chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca)

INTERVENTIONS:
Biological: H9N2 (6-2) AA ca Reassortant (A/chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca) — Live attenuated H9N2 (6-2) AA ca Reassortant (A/chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca) vaccine

SUMMARY:
Avian influenza (AI), or bird flu, has recently become a major health concern in Asia and other parts of the world. The purpose of this study is to test the safety of and immune response to a new AI vaccine in healthy adults.

Study hypothesis: Influenza A viruses are widely distributed in nature and infect a wide variety of birds and mammals. The direct transmission of avian influenza viruses from birds to humans has recently become a major health concern in Asia and other parts of the world, raising concern of a possible influenza pandemic in humans. This vaccine will evaluate the safety, infectivity and immunogenicity of Live Influenza A vaccine H9N2 (6-2) AA ca reassortant (A/chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca), a cold-adapted, live attenuated virus vaccine administered intranasally for the protection of humans against pandemic influenza viruses of the H9N2 subtype.

DETAILED DESCRIPTION:
AI viruses in their natural reservoir in waterfowl are the source from which novel HA and NA subtypes are introduced into the human population, and have the potential to initiate an influenza pandemic. This study will evaluate the safety and immunogenicity of a live, attenuated, cold-adapted reassortant AI virus vaccine, H9N2 (6-2) AA ca Reassortant (A/chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca).

Patient participation in this study will be for at least 60 days, with patients followed for at least 42 days after vaccination. In this study, participants will be enrolled sequentially, from highest to lowest dose of vaccine, into one of three groups. At study entry at Day 0, participants will be admitted to the hospital in order to familiarize them with trial procedures. Blood and nasal wash samples will be collected prior to vaccination. On Day 2, participants will have a physical exam and will receive one dose of vaccine; the vaccine will be administered as nose drops. Participants will undergo directed physical examinations daily while they are in the hospital. Nasal washes will also be collected daily from the day of admission through the day prior to discharge to test for the presence of vaccine virus. Participants may be discharged from the hospital after 3 consecutive negative viral cultures, but not before Day 14. Additional blood collection will occur daily from Day 0 to Day 7 and again on Day 21. Participants will return for follow-up visits 28 to 32 days and 42 to 46 days after receiving the vaccine. Blood and nasal wash collection will occur at these 2 study visits, and participants will also have directed physical exams.

Depending on the immune response to the first dose of vaccine, some participants may be asked to return to the hospital 1 to 2 months after their first vaccination to receive an additional dose of vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Born after 1968
* Good general health
* Available for the duration of the trial

Exclusion Criteria:

* Clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the ability of the volunteer to understand and cooperate with the study
* Liver, renal, or hematologic disease
* Alcohol or drug abuse within 12 months of study entry
* History of severe allergic reaction or anaphylaxis
* Current asthma or reactive airway disease
* History of Guillain-Barre syndrome
* HIV-1 infected
* Hepatitis C virus infected
* Positive for hepatitis B surface antigen (HBsAg)
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs within 30 days of study entry. Participants who have used topical corticosteroids are not excluded.
* Live vaccine within 4 weeks of study entry
* Killed vaccine within 2 weeks of study entry
* Absence of spleen
* Blood products within 6 months of study entry
* Current smoker
* Have traveled to the Southern Hemisphere or Asia within 30 days prior to study entry
* Have traveled on a cruise ship within 30 days prior to study entry
* Work in the poultry industry
* Investigational agents within 60 days prior to study entry, or currently participating in another investigational vaccine or drug trial
* Allergy to eggs or egg products
* Purified protein derivative (PPD) positive (positive tuberculosis [TB] test)
* Family member with immunodeficiency
* Other condition that, in the opinion of the investigator, would affect the participant's participation in the study
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-06; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events and other adverse effects for each dose of the H9N2 G9/AA ca reassortant vaccine | Throughout study
Immunogenicity and infectivity for each dose of the H9N2 G9/AA ca reassortant vaccine | Throughout study

SECONDARY OUTCOMES:
To compare antibody responses | At Days 28 and 42
To determine the number of vaccinees infected with the H9N2 G9/AA ca reassortant vaccine candidate. | Throughout study
If 10^7 , 10^5 , and 10^3 TCID50 doses of vaccine are administered, to compare the infectivity rates, safety, and immunogenicity between dose groups, and to estimate the HID50 for this vaccine | Throughout study
To determine the phenotypic stability of vaccine virus shed | Throughout study
To determine whether immunogenicity is enhanced by a second dose of vaccine, and whether the first dose of vaccine restricts replication of the second dose | At study completion
To evaluate T-cell mediated and innate immune responses against the H9N2 G9/AA ca reassortant vaccine candidate | Throughout study
To develop a serum bank so that the capacity of the H9N2 G9/AA ca reassortant vaccine candidate to elicit HI and neutralizing antibodies to future H9N2 influenza viruses can be tested | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Center of Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Chen H, Matsuoka Y, Swayne D, Chen Q, Cox NJ, Murphy BR, Subbarao K. Generation and characterization of a cold-adapted influenza A H9N2 reassortant as a live pandemic influenza virus vaccine candidate. Vaccine. 2003 Oct 1;21(27-30):4430-6. doi: 10.1016/s0264-410x(03)00430-4. PMID 14505926
- [Background] Choi YK, Ozaki H, Webby RJ, Webster RG, Peiris JS, Poon L, Butt C, Leung YH, Guan Y. Continuing evolution of H9N2 influenza viruses in Southeastern China. J Virol. 2004 Aug;78(16):8609-14. doi: 10.1128/JVI.78.16.8609-8614.2004. PMID 15280470
- [Background] Stephenson I, Nicholson KG, Wood JM, Zambon MC, Katz JM. Confronting the avian influenza threat: vaccine development for a potential pandemic. Lancet Infect Dis. 2004 Aug;4(8):499-509. doi: 10.1016/S1473-3099(04)01105-3. PMID 15288823
- [Background] Swayne DE. Vaccines for List A poultry diseases: emphasis on avian influenza. Dev Biol (Basel). 2003;114:201-12. PMID 14677690
- [Derived] Karron RA, Callahan K, Luke C, Thumar B, McAuliffe J, Schappell E, Joseph T, Coelingh K, Jin H, Kemble G, Murphy BR, Subbarao K. A live attenuated H9N2 influenza vaccine is well tolerated and immunogenic in healthy adults. J Infect Dis. 2009 Mar 1;199(5):711-6. doi: 10.1086/596558. PMID 19210163